CLINICAL TRIAL: NCT05733624
Title: A Multicenter, Active Control, Parallel Group, Randomized, Double-blind, Phase II Clinical Trial to Evaluate the Efficacy and Safety of SCAI-001 Eye Drops in Patients With Dry Eye Disease
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of SCAI-001 Compared to Restasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCAI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCAI-001-201
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye; Cyclosporine
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions; Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SCAI-001 0.01% (Experimental): Cyclosporine 0.01%
  Interventions: Drug: SCAI-001 0.01% eyedrop
- SCAI-001 0.02% (Experimental): Cyclosporine 0.02%
  Interventions: Drug: SCAI-001 0.02% eyedrop
- Restasis (Active Comparator): Cyclosporine 0.05%
  Interventions: Drug: Restasis 0.05% eyedrop

INTERVENTIONS:
Drug: SCAI-001 0.01% eyedrop — BID for 12weeks
  Other Names: Cyclosporine 0.01%
  Arms: SCAI-001 0.01%
Drug: SCAI-001 0.02% eyedrop — BID for 12weeks
  Other Names: Cyclosporine 0.02%
  Arms: SCAI-001 0.02%
Drug: Restasis 0.05% eyedrop — BID for 12weeks
  Other Names: Cyclosporine 0.05%
  Arms: Restasis

SUMMARY:
This study is planned to Evaluate the Efficacy and Safety of SCAI-001 Eye Drops(Cyclosporine 0.01%, 0.02%) compared to Restasis(Cyclosporine 0.05%) in Patients with Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female who over 19 years old
2. Those who have dry eye symptoms (Dryness, Grittiness, soreness, irritation, watering, etc.)
3. Those who meet below criteria at least one of two eyes;

   * Those who have over than score 2 in corneal staining test-Oxford grading
   * Tear secretion test without anesthesia(Schirmer test) result would be under 10mm/5min (If the test result is 0mm/5min, it should be over than 3mm/5min on the nasal stimulation schirmer test in the same eye)
   * TBUT(Tear film break-up time) test result should be under 10sec.
4. The corrected visual acuity is 0.2 or more.

Exclusion Criteria:

1. Those who have clinically significant eye disease not related to dry eye syndrome
2. Those who are in medication of systemic steroid or immunosuppressant 90days before screening visit
3. Those who have worn contact lenses before 72hours or have to wear contact lenses or disagree not to wear contact lenses during study period
4. Those who have medical history with intraocular surgery 12months before screening visit
5. Those who have diagnosed with glaucoma or have an intraocular pressure over than 21mmHg at least in one of the eyes
6. Those who have medicated cyclosporine eye-drops 6weeks before screening visit
7. Those who have underwent any eye correction surgery such as LASIK(Laser-assistant in situ keratomileusis) 12 months before screening visit
8. Those who have underwent a silicone lacrimal punctal occlusion or cauterization of the punctum excluding collagen lacrimal punctal occlusion 90 days before screening visit
9. Those who have received other investigational drugs/devices 30 days before screening visit
10. Those who are inappropriate for participating in this study according to investigator's judgement

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Tear volume | Change from baseline at 12 weeks
  Schirmer's test

SECONDARY OUTCOMES:
Tear volume | Change from baseline at 4, 8 weeks
  Schirmer's test
Corneal staining score with fluorescein | Change from baseline at 4, 8, 12 weeks
  Oxford grading
conjunctival staining score with Lissamine green | Change from baseline at 4, 8, 12 weeks
  Oxford grading
Tear film break-up time | Change from baseline at 4, 8, 12 weeks
  Measured three times and recorded up to 1/100
Standard patient evaluation of eye dryness questionnaire | Change from baseline at 4, 8, 12 weeks
  written by the subject
Ocular surface disease index | Change from baseline at 4, 8, 12 weeks
  written by the subject
Total number of rescue medication used | 12weeks
  sourced by patient diary

CONTACTS AND LOCATIONS:
Overall Officials: Lee, MD, PhD, Principal Investigator — Pusan National Univ. Hospital
Locations (11):
- South Korea (11):
  - The Catholic University of korea, Bucheon ST.Mary's Hospital, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Pusan National Univ. Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Asan Medical Center, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No